CLINICAL TRIAL: NCT00419770
Title: The Deferasirox-AmBisome Therapy for Mucormycosis (DEFEAT Mucor) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Gilead Sciences (Industry); Astellas Pharma Inc (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12842
Record Dates: First submitted 2007-01-05; First posted 2007-01-09 (Estimated); Results first posted 2011-10-06 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Mucormycosis
Keywords: zygomycosis; Rhizopus; iron; iron-chelation; adjunctive therapy
MeSH Terms: conditions — Mucormycosis; Zygomycosis | interventions — Deferasirox; liposomal amphotericin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): Deferasirox
  Interventions: Drug: deferasirox; Drug: Liposomal amphotericin B
- A (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Liposomal amphotericin B

INTERVENTIONS:
Drug: deferasirox — 20 mg/kg enterally per day
  Other Names: Exjade
  Arms: B
Drug: Placebo
  Arms: A
Drug: Liposomal amphotericin B

SUMMARY:
The purpose of this study is to determine if the addition of the medication, deferasirox, to standard antifungal therapy for the infection, mucormycosis, is safe and effective

DETAILED DESCRIPTION:
Because of its extremely high morbidity and mortality, it is imperative to look for new antifungal therapies to treat mucormycosis. The agents of mucormycosis are exquisitely sensitive to iron availability, and we and others have demonstrated that iron chelation therapy improves the survival of rodents with mucormycosis. Deferasirox (Exjade) is the first orally bioavailable iron chelator approved for use in the United States (US) by the Food and Drug Administration (FDA), with an indication for treatment of iron overload from chronic transfusions. In clinical studies, deferasirox has been well tolerated and effective in iron-overloaded patients.

Although the safety and efficacy of deferasirox have been extensively evaluated in iron-overloaded patients, there are minimal data in non-iron-overloaded patients or in infected patients. Therefore, the safety and efficacy of deferasirox in patients with mucormycosis is unclear, and confirming safety in the current study, at the currently planned dose, is required to lay the groundwork for a future phase III clinical trial.

This is a prospective, phase II, randomized, double-blinded, placebo-controlled study of liposomal amphotericin B (LAmB; AmBisome) plus deferasirox vs. LAmB plus placebo for mucormycosis infection. Twenty patients with proven or probable mucormycosis (except for isolated skin infection) by consensus EORTC/MSG criteria, who have received less than 14 days of antifungal therapy for mucormycosis, and who have had radiographic imaging by CT or MRI within the past 72 hours that shows evidence of infection, will be randomized to receive LAmB plus deferasirox or placebo (n = 10 per arm), with randomization stratified by study site.

The primary objective is to determine the safety and tolerability of adjunctive deferasirox therapy in patients being treated with LAmB for mucormycosis, and to obtain exploratory data on the efficacy of the iron chelation treatment. The exploratory efficacy endpoint will be the global response rate (composite of clinical and radiographic response) at end of study drug administration, as determined by a blinded adjudication committee.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 2 years.
* Proven or probable invasive mucormycosis, as defined by modification of consensus European Organization for Research and Treatment of Cancer (EORTC)/Mycosis Study Group (MSG) criteria. In brief, proven mucormycosis is defined as: 1) histopathologic or cytopathologic examination showing broad-based, aseptate, ribbon-like hyphae consistent with Mucorales from needle aspiration or biopsy specimen, with evidence of associated tissue damage (either microscopically or unequivocally by imaging); OR 2) a positive culture result for a sample obtained by sterile procedure from normally sterile and clinically or radiologically abnormal site consistent with infection, excluding urine and mucous membranes. Probable mucormycosis is defined as: 1) an at-risk host; AND 2) positive culture, cytology, or polymerase chain reaction (PCR) test (run at a CLIA-certified clinical microbiology laboratory) from sputum, bronchoalveolar lavage (BAL), endoscopy/colonoscopy, or sinus aspirate/biopsy; AND 3) 1 major or 2 minor clinical criteria.
* Radiographic study by Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) has been obtained within 4 calendar days prior to enrollment and shows evidence of infection (i.e. focal nodule, mass, or abscess, or enhancement, or evidence of tissue edema or destruction that is not attributed to post-surgical reaction).
* Subject or authorized decision maker able to provide informed consent.

Exclusion Criteria:

* High likelihood of death within the 48 h after enrollment (investigator's discretion).
* High likelihood of death due to factors unrelated to mucormycosis (e.g. due to uncontrolled and/or relapsed malignancy, severe graft versus host disease, other underlying diseases, etc.) within 30 days following enrollment (investigator's discretion).
* Patient unable to receive enteral medication (oral or via feeding tube).
* Infection limited to the supra-fascial skin (skin lesions in the presence of disseminated disease, deep invasive tissue infection spreading from a primary skin site, or subcutaneous infections extending to fascia are allowed).
* Patient has received > 14 days of polyene antifungal therapy (i.e. amphotericin B deoxycholate, liposomal amphotericin B, amphotericin B lipid complex, or amphotericin B colloidal dispersion) at the time of screening.
* Patient is already taking deferasirox therapy for any reason at the time of screening.
* Patient is allergic to or intolerant of deferasirox or LAmB.
* Patient has significant renal dysfunction at the time of screening, defined as serum creatinine of > 3 mg/dL or a calculated creatinine clearance of < 30 ml/min (by the Cockroft-Gault formula: (140 - age (yrs) * wt (kg)) * 0.85 (for females) / (72 * serum creatinine (mg/dL)).
* Patient has significant hepatic dysfunction at the time of screening, defined as BOTH an AST or ALT > 10 times the upper limit of normal, AND a direct (not total) bilirubin > 5 times the upper limit of normal.
* Women of child-bearing potential (those with menses within the last year) with a positive serum pregnancy test.
* Enrollment refused by the primary physician.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Spellberg, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - UCSF, San Francisco, California
  - University of Miami, Miami, Florida
  - Duke University, Durham, North Carolina
  - Summa Health Systems, Akron, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Spellberg B, Edwards J Jr, Ibrahim A. Novel perspectives on mucormycosis: pathophysiology, presentation, and management. Clin Microbiol Rev. 2005 Jul;18(3):556-69. doi: 10.1128/CMR.18.3.556-569.2005. PMID 16020690
- [Background] Ibrahim AS, Edwards JE Jr, Fu Y, Spellberg B. Deferiprone iron chelation as a novel therapy for experimental mucormycosis. J Antimicrob Chemother. 2006 Nov;58(5):1070-3. doi: 10.1093/jac/dkl350. Epub 2006 Aug 23. PMID 16928702
- [Background] Reed C, Ibrahim A, Edwards JE Jr, Walot I, Spellberg B. Deferasirox, an iron-chelating agent, as salvage therapy for rhinocerebral mucormycosis. Antimicrob Agents Chemother. 2006 Nov;50(11):3968-9. doi: 10.1128/AAC.01065-06. Epub 2006 Sep 25. No abstract available. PMID 17000743
- [Background] Boelaert JR, Van Cutsem J, de Locht M, Schneider YJ, Crichton RR. Deferoxamine augments growth and pathogenicity of Rhizopus, while hydroxypyridinone chelators have no effect. Kidney Int. 1994 Mar;45(3):667-71. doi: 10.1038/ki.1994.89. PMID 8196268
- [Derived] Spellberg B, Ibrahim AS, Chin-Hong PV, Kontoyiannis DP, Morris MI, Perfect JR, Fredricks D, Brass EP. The Deferasirox-AmBisome Therapy for Mucormycosis (DEFEAT Mucor) study: a randomized, double-blinded, placebo-controlled trial. J Antimicrob Chemother. 2012 Mar;67(3):715-22. doi: 10.1093/jac/dkr375. Epub 2011 Sep 20. PMID 21937481

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferasirox: Deferasirox (20 mg/kg/d for 14 days) plus liposomal amphotericin (minimum dose of 5 mg/kg thrice weekly)
- Placebo: Placebo control plus background liposomal amphotericin
Period: Overall Study
Arm/Group | Deferasirox | Placebo
Started | 11 | 9
Completed | 6 | 8
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Deferasirox: Deferasirox plus liposomal amphotericin
- Total: Total of all reporting groups
Arm/Group | Deferasirox | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 3 | 2 | 5
Age, Continuous [Median (Full Range); unit: years] | 59 [30 to 71] | 47 [40 to 75] | 52 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Adjunctive Deferasirox Therapy in Patients Being Treated With LAmB for Mucormycosis
Time Frame: 14 days
Reporting Status: Not Posted

2. Primary Outcome: Global Response Rate (Composite of Clinical and Radiographic Response) at End of Study Drug Administration, as Determined by a Blinded Adjudication Committee
Time Frame: 14 days
Reporting Status: Not Posted

3. Secondary Outcome: Deferasirox Pharmacokinetic and Pharmacodynamic Parameters
Time Frame: 7 days
Reporting Status: Not Posted

4. Secondary Outcome: Survival, Radiographic Improvement, Clinical Response, Time to Survival, Deferasirox vs. Free Iron Level Correlation
Time Frame: Up to 90 days
Reporting Status: Not Posted

5. Primary Outcome: Total Adverse Events
Time Frame: 30 Days After End of Therapy
Measure: Number; unit: Events
Arm/Group | Deferasirox | Placebo
Number analyzed (Participants) | 11 | 9
Events | 16 | 16

ADVERSE EVENTS:
Arm/Group | Deferasirox | Placebo
Serious Adverse Events (participants affected / at risk) | 8/11 | 4/9
Other Adverse Events (participants affected / at risk) | 8/11 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (N=11) | Placebo (N=9)
Progressive Infection (Infections and infestations) | 1 (1) | 0 (0)
Progression of underlying disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Respiratory Failure (General disorders) | 2 (2) | 2 (2)
Renal Failure (General disorders) | 1 (1) | 0 (0)
Liver failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting/interolerance of study drug (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intracranial bleeding (Nervous system disorders) | 1 (1) | 0 (0)
arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
alveolar hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
bacterial pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (N=11) | Placebo (N=9)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Exophthalmos (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurry vision (Eye disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte abnormalities (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Myoclonus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 0 (0) | 2 (3)
Respiratory distress (General disorders) | 1 (1) | 0 (0)
Rash (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No